CLINICAL TRIAL: NCT00726128
Title: A Multi-Center Prospective Patient Outcomes Evaluation of the EBI Vuelock™ Anterior Cervical Plate System
Brief Title: Patient Outcomes Evaluation of the EBI Vuelock™ Anterior Cervical Plate System
Acronym: VueLock
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-005-04
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Trauma; Tumor; Pseudarthrosis; Scoliosis; Degenerative Disc Disease
Keywords: Degenerative Disc disease (DDD)
MeSH Terms: conditions — Wounds and Injuries; Neoplasms; Pseudarthrosis; Scoliosis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VueLock™ Anterior Cervical Plate Group: VueLock™ Anterior Cervical Plate, Implanted in subjects having an ACDF (Anterior cervical discectomy and fusion)
  Interventions: Device: VueLock™ Anterior Cervical Plate

INTERVENTIONS:
Device: VueLock™ Anterior Cervical Plate — Implanted in subjects having an ACDF (Anterior cervical discectomy and fusion)

SUMMARY:
To prospectively collect radiographic and outcome data on patients who are having cervical spine fusion surgery with the VueLock™ Anterior Cervical Plate System

DETAILED DESCRIPTION:
The purpose is to prospectively collect radiographic and outcome data on patients who are having cervical spine fusion surgery with the VueLock™ Anterior Cervical Plate System.

ELIGIBILITY:
Inclusion Criteria:

1. The patient will undergo anterior cervical fusion with the VueLock™ Anterior Cervical Plate System for treatment of degenerative disc disease (as defined by neck pain of discogenic origin of the disc confirmed by patient history and radiographic studies), trauma, tumors, deformity (defined as kyphosis, lordosis, or scoliosis), pseudarthrosis, and/or failed previous fusion.
2. The patient must be available for follow-up during the study.
3. The patient must be skeletally mature (epiphyses closed).

Exclusion Criteria:

1. Patients with other pathology at the involved spinal level, e.g., osteomyelitis, Paget's disease, pathologic fracture, etc.
2. Patients with a disease entity or condition that totally precludes the possibility of bony fusion such as known active cancer, etc.
3. Pregnant or nursing females.
4. Patients who in the opinion of the investigator would be psychologically unwilling or unable to understand or complete the protocol, especially those unwilling or unstable to participate in the follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects from multiple centers with disease of the cervical spine
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 1998-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients with radiographic fusion | 24 Months

SECONDARY OUTCOMES:
Neck Disability Index and Short Form Health Survey (SF-36) scores, change from baseline | 24 Month

CONTACTS AND LOCATIONS:
Overall Officials: John Evangelsita, MD, Study Chair — EBI, LLC dba Biomet Spine, Biomet Trauma, Biomet Osteobiologics and Biomet Bracing
Locations (4):
- United States (4):
  - Palo Alto Medical Foundation, Palo Alto, California
  - Alvarado Orthopedic Clinic, San Diego, California
  - American health Network, Avon, Indiana
  - Raliegh Orthopedic Research Foundation, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided